CLINICAL TRIAL: NCT03102957
Title: Cartography of Functional and Epileptic Cerebral Areas by Functional MRI and Electroencephalography in Epileptic Patients Before and After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC09.21
Record Dates: First submitted 2017-03-22; First posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: 2 arms : epileptic patient and healthy volonteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- epileptic patients (Experimental): 2 functional MRI (pre and post resective surgery) with memory and language tasks
  Interventions: Other: functional MRI
- Healthy volunteers (Other): 1 functional MRI with memory and language tasks
  Interventions: Other: functional MRI

INTERVENTIONS:
Other: functional MRI

SUMMARY:
Exploring the reorganization (plasticity) of neuroanatomic networks associated with language and memory in patients with left (or dominant hemisphere) temporal lobe epilepsy using functional MRI (fMRI)

DETAILED DESCRIPTION:
The purpose of this study is to explore the reorganization of neuroanatomic networks associated with language and memory in adult patients with temporal lobe epilepsy (ELT). By using functional MRI, patients will be examined before and after surgery. Cerebral plasticity, defined in terms of intrinsic variables such as the topography of the activated regions, will be explored according to some extrinsic factors such as the age at onset of crises (before or after 5-6 years), whether or not Hippocampal sclerosis, hemispheric predominance of language (left or right).

ELIGIBILITY:
Inclusion Criteria:

* epileptic patients
* medical exam before inclusion
* social security affiliation
* Pharmaco-resistant epilepsy

Exclusion Criteria:

* MRI contraindication
* pregnant women
* breastfeeding mothers
* person under tutorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-06-17 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
neuronal reorganization exploration in language and memory area thanks to functionnal MRI | one hour for each exam
  fMRI exam before and after resection surgery of epileptogenic area: assess (plasticity) of neuroanatomic networks associated with language and memory - examined before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre KRAINIK, PhD, Principal Investigator — University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No